## Statistical Analysis Plan January 30, 2019

Survey providers from Internal Medicine (IM) and Family Medicine (FM) to evaluate fall treatment. Educate providers on new protocol. Survey results will be analyzed and used to develop to develop educational care protocol for treatment which will be communicated to providers at grand rounds.

Twelve months after grand rounds, a second survey of IM and FM providers will be conducted to determine how well physical therapy referrals and Vitamin D supplementation dosages aligned with the established protocol.

Associations between pre/post results for categorical variables will be tested with chi-square or Fisher's Exact test.

For comparisons of means for Likert variables, a two sample t-test will be used.

Statistical analysis will be completed using R statistical software program. R Core Team (2019). R: A language and environment for statistical computing. R Foundation for Statistical Computing, Vienna, Austria. URL https://www.R-project.org/.

Statistical significance is defined as a p value of 0.05 or less.